CLINICAL TRIAL: NCT04338698
Title: Pakistan Randomized and Observational Trial to Evaluate Coronavirus Treatment
Brief Title: Hydroxychloroquine, Oseltamivir and Azithromycin for the Treatment of COVID-19 Infection: An RCT
Acronym: PROTECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shehnoor Azhar (Other)
Responsible Party: Sponsor-Investigator, Shehnoor Azhar, Study Coordinator, University of Health Sciences Lahore
Organization: University of Health Sciences Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12(06)/2016-Coord
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Oseltamivir; Azithromycin

STUDY DESIGN:
Intervention Model Description: Adaptive design (sample size given below is indicative)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Control Intervention (Active Comparator): Hydroxychloroquine
  Interventions: Drug: Hydroxychloroquine
- Comparator 1 (Experimental): Azithromycin
  Interventions: Drug: Azithromycin
- Comparator 2 (Experimental): Oseltamivir
  Interventions: Drug: Oseltamivir
- Comparator 3 (Experimental): Hydroxychloroquine + Azithromycin
  Interventions: Drug: Hydroxychloroquine; Drug: Azithromycin
- Comparator 4 (Experimental): Hydroxychloroquine + Oseltamivir
  Interventions: Drug: Hydroxychloroquine; Drug: Oseltamivir
- Comparator 5 (Experimental): Oseltamivir + Azithromycin
  Interventions: Drug: Oseltamivir; Drug: Azithromycin
- Comparator 6 (Experimental): Hydroxyquinine + Oseltamivir + Azithromycin
  Interventions: Drug: Hydroxychloroquine; Drug: Oseltamivir; Drug: Azithromycin
- Observational Cohort (No Intervention): Non-consenting to randomization

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine Sulfate (200 mg orally thrice a day for 5 days)
  Arms: Comparator 3; Comparator 4; Comparator 6; Control Intervention
Drug: Oseltamivir — Oseltamivir (75 mg orally twice a day for 5 days)
  Arms: Comparator 2; Comparator 4; Comparator 5; Comparator 6
Drug: Azithromycin — Azithromycin (500 mg orally once a day on day 1, followed by 250 mg orally daily on days 2-5)
  Arms: Comparator 1; Comparator 3; Comparator 5; Comparator 6

SUMMARY:
To evaluate the effectiveness of Hydroxychloroquine Sulfate (200 mg orally 8hr thrice a day for 5 days) vs oseltamivir (75 mg orally twice a day for 5 days) vs Azithromycin (500 mg orally daily on day 1, followed by 250 mg orally twice a day on days 2-5) alone and in combination (in all seven groups), in clearing the coronavirus nucleic acid from throat and nasal swab and in bringing about clinical improvement on day 7 of follow-up (primary outcomes).

DETAILED DESCRIPTION:
A scientific taskforce notified by the Ministry of Science and Technology of the Government of Pakistan will oversee a comprehensive cohort study. Within this cohort, a multicenter, adaptive, randomized controlled trial will evaluate, among eligible SARS-Cov-2 (COVID-19) infected patients receiving standard supportive care who consent to randomization following a new diagnosis in Pakistan, if Hydroxychloroquine Sulfate alone (control intervention) vs a series of alternatives (comparator interventions) including Oseltamivir and Azithromycin alone and in combination with Hydroxychloroquine Sulfate is effective in clearing the coronavirus and improving the clinical course of the disease. Those not consenting to randomization will be followed up for outcomes of SARS-Cov-2 infection with supportive care only. Findings of this study are expected to inform clinical care and public health protocols and policies for management of SARS-Cov-2.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed SARS-CoV-2 (COVID-19) infection by a positive test result
2. Either gender
3. Symptomatic for example fever, dry Cough, difficulty to breathe

Exclusion Criteria:

1. Confirmed absence of SARS-CoV-2 (COVID-19) infection by a negative test result
2. Have chronic conditions such as heart disease, liver and kidney failure
3. Pregnant or currently lactating
4. Immunocompromise and/or systemic disease(s)
5. On other antiviral drugs
6. History of allergy to any of the drugs to be administered in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-22 (Actual)

PRIMARY OUTCOMES:
Laboratory Result | Day 07 on follow-up
  The laboratory-based primary outcome will be turning test negative for COVID-19 on RT-qPCR calculated as viral load of < 150 i.u
Clinical Outcome | Day 07 on follow-up
  The clinical primary outcome will be improvement of two points on a seven-category ordinal scale shown below:
  1. Not hospitalized, able to resume normal activities
  2. Not hospitalized, but unable to resume normal activities
  3. Hospitalization, not requiring supplemental oxygen
  4. Hospitalization, requiring supplemental oxygen
  5. Hospitalization, requiring noninvasive mechanical ventilation
  6. Hospitalization, requiring invasive mechanical ventilation
  7. Death

CONTACTS AND LOCATIONS:
Overall Officials: Javed Akram, FRCP, Principal Investigator — University of Health Sciences Lahore
Locations (11):
- Pakistan (11):
  - Nawaz Sharif Medical College, Dhok Gujra
  - Faislabad Medical University, Faisalābad
  - Gujranwala Medical College, Gujranwala
  - Szabmu-Pims, Islamabad
  - Akram Medical Complex, Lahore
  - Fatima Jinnah Medical University, Lahore
  - King Edward Medical University-Mayo Hospital, Lahore
  - Lahore General Hospital, Lahore
  - Khyber Teaching Hospital, Peshawar
  - Rawalpindi Medical University, Rawalpindi
  - Sargodha Medical College, Sargodha

IPD SHARING:
Plan to Share IPD: Yes
On completion of study, investigators are open to participation in planned IPD projects with a prospective registration, subject to appropriate approvals

REFERENCES:
- [Derived] Azhar S, Akram J, Latif W, Ibanez NC, Mumtaz S, Rafi A, Aftab U, Iqtadar S, Shahzad M, Syed F, Zafar B, Fatima N, Afridi SS, Akram SJ, Chaudhary MA, Sadiq F, Goraya S, Hanif M, Ashraf V, Ashraf S, Akram H, Khaliq T. Effectiveness of early pharmaceutical interventions in symptomatic COVID-19 patients: A randomized clinical trial. Pak J Med Sci. 2024 May-Jun;40(5):800-810. doi: 10.12669/pjms.40.5.8757. PMID 38827854
- [Derived] Azhar S, Akram J, Shahzad M, Latif W, Khan KS. Protocol of Pakistan randomized and observational trial to evaluate coronavirus treatment among newly diagnosed patients with COVID-19: Azithromycin, Oseltamivir, and Hydroxychloquine. Pak J Med Sci. 2022 May-Jun;38(5):1401-1408. doi: 10.12669/pjms.38.5.5512. PMID 35799756
- [Derived] Akram J, Azhar S, Shahzad M, Latif W, Khan KS. Pakistan Randomized and Observational Trial to Evaluate Coronavirus Treatment (PROTECT) of Hydroxychloroquine, Oseltamivir and Azithromycin to treat newly diagnosed patients with COVID-19 infection who have no comorbidities like diabetes mellitus: A structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Aug 8;21(1):702. doi: 10.1186/s13063-020-04616-4. PMID 32771032